CLINICAL TRIAL: NCT06083857
Title: An Open-Label Phase I/II Study to Evaluate the Safety and prelimiBasnary Efficacy of Amivantamab and Tepotinib Combination in MET-altered Non-small Cell Lung Cancer (NSCLC)
Brief Title: PhI/II Study of Amivantamab and Tepotinib Combo in MET-altered Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0860; NCI-2023-08689 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Amivantamab and Tepotinib Combination (Experimental): Participants will be given 2 investigational drugs (amivantamab and tepotinib) and come to the clinic for study visits every 4 weeks.
  Interventions: Drug: Amivantamab; Drug: Tepotinib

INTERVENTIONS:
Drug: Amivantamab — Given by IV (vein)
Drug: Tepotinib — Given by PO

SUMMARY:
To learn if the combination of amivantamab and tepotinib can help to control NSCLC. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

1. For the safety run-in portion of the trial:
2. To evaluate dose-limiting toxicity (DLT) and to establish the recommended phase II dose (RP2D) of amivantmab given in combination with tepotinib in patients with advanced MET-altered NSCLC. The primary endpoint is dose-limiting toxicity (DLT) and recommended phase 2 dose (RP2D).
3. For the efficacy portion of the trial:
4. To preliminarily assess efficacy of amivantamab + tepotinib combination in cohort A (MET exon 14 skipping TKI-naïve) , in terms of objective response rate.

Secondary Objectives

1. Determine whether amivantamab + tepotinib improves objective response rate in each cohort (cohort B and cohort C)
2. Determine whether amivantamab + tepotinib improves disease control rate (DCR) in each cohort
3. Determine whether amivantamab + tepotinib improves Duration of Response (DoR) in each cohort
4. Determine the safety and tolerability of amivantamab + tepotinib in each cohort

Exploratory Objectives

1. Explore the association of baseline genomic profiles (from tumor, germline DNA, and ctDNA) with clinical benefit in patients treated with amivantamab + tepotinib
2. Explore resistance mechanisms to amivantamab + tepotinib combination. At the time of progression, patients will undergo ctDNA genomic tests and a biopsy (optional). The purpose of this additional tissue acquisition is for molecular analysis and comparison with the initial specimen, to determine if there are changes in molecular alterations or pathways that shed light on mechanisms of resistance.
3. Determine the immunomodulatory effects of amivantamab + tepotinib combination.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health inf ormation prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Histologically or cytologically confirmed non-small cell lung cancer.
4. Locally advanced or metastatic disease, not amenable to curative surgery or radiotherapy.
5. Patients must have one of the following:

   * NSCLC which harbors MET Exon 14 skipping alterations detected in the tissue or ctDNA (safety cohort and cohort A [MET ex14 TKI-naïve] and B [MET ex14 TKI-refractory])
   * MET gene amplification determined in tissue by next-generation sequencing (NGS) as copy-number gain (CNG>=10) or FISH assay (MET:CEP7>=2.0) (safety cohort and cohort C [MET amplification or overexpression cohort]
   * MET gene amplification determined in ctDNA (definition of gain per ctDNA testing platform) (safety cohort and cohort C [MET amplification or overexpression cohort]
   * MET overexpression by IHC 3+ (safety cohort and cohort C [MET amplification or overexpression cohort]
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Measurable disease per RECIST 1.1.
8. Patients with brain metastases are eligible if they are asymptomatic, are treated, or are neurologically stable for at least two weeks without the use of steroids or on stable or decreasing dose of ≤ 15 mg daily prednisone (or equivalent).
9. Ability to take pills by mouth.
10. Previous treatment with cytotoxic chemotherapy or immunotherapy is allowed.
11. Patients must have adequate bone marrow and organ functions.

    * Hemoglobin ≥10 g/dL
    * ANC ≥1.5 x 109 /L
    * Platelets ≥75 x 10 9 /L
    * AST and ALT ≤3 x ULN
    * Total bilirubin ≤1.5 x ULN; subjects with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits
    * Serum creatinine <1.5 x ULN or if available, calculated or measured creatinine clearance >50 mL/min/1.73 m2 ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal
12. A woman of childbearing potential must have a negative serum pregnancy test at screening and within 7 days of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.
13. A woman must be compliant with the Contraceptive Guidance and Collection of Pregnancy Information:

    1. Not of childbearing potential
    2. Of child-bearing potential and practicing true abstinence during the entire period of the study, including up to 6 months after the last dose of study treatment is given
    3. Of childbearing potential and practicing 2 methods of contraception, including 1 highly effective user independent method and a second method.

    Participant must agree to continue contraception throughout the study and through 6 months after the last dose of study treatment.

    • Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) the woman must begin birth control, as described above.
14. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study treatment.
15. A man must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 6 months after receiving the last dose of study treatment. A man who is sexually active with a woman of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and his partner must also be practicing a highly effective method of contraception (ie, established use of oral, injected, or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]).

    If the participant is vasectomized, he must still use a condom (with or without spermicide) for prevention of passage of exposure through ejaculation, but his female partner is not required to use contraception.
16. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment.
17. Participant must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

1. For cohort A (METex14 TKI-naïve only), prior targeted therapy to c-MET is not allowed, which includes small molecule TKIs, such as tepotinib, capmatinib, savolitinib, or crizotinib. Prior amivantamab is also not allowed.
2. Patients whose tumor harbors other oncogene-driver mutations, such as EGFR mutation, KRASG12C mutation, ALK-fusion, with prior targeted therapies, such as osimertinib, sotorasib, and other TKI, are not allowed.
3. Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) Note: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.
4. Positive hepatitis C antibody (anti-HCV). Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
5. Other clinically active or chronic liver disease.
6. Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

   * Receiving ART that may interfere with study treatment (consult with Principal Investigator for review of medication prior to enrollment)
   * CD4 count <350 at screening
   * AIDS-defining opportunistic infection within 6 months of start of screening
   * Not agreeing to start ART and be on ART>4 weeks plus having HIV viral load <400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV controlled).
7. Participant has active cardiovascular disease including, but not limited to:

   * A medical history of deep vein thrombosis or pulmonary embolism within 1 month prior to first dose of study drug or any of the following within 6 months prior to the first dose of study drug: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, uncontrolled hypertension, clinically significant cardiac arrythmia, or any acute coronary syndrome. Clinically non-significant thrombosis, such as non-obstructive catheter-associated clots, incidental or asymptomatic pulmonary embolism, are not exclusionary.
   * Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalization for CHF (any NYHA class; refer to Appendix: New York Heart Association Criteria) within 6 months of study Day 1.
8. Subject has uncontrolled inter-current illness, including but not limited to poorly controlled diabetes, ongoing or active infection (i.e., has discontinued all antibiotics for at least one week prior to first dose of study drug), or psychiatric illness/social situation that would limit compliance with study requirements. Subjects with medical conditions requiring chronic continuous oxygen therapy are excluded.
9. Any ophthalmologic condition that is clinically unstable (consult with Principal Investigator for review of the condition prior to enrollment).
10. Participant has an active or past medical history of ILD/pneumonitis, including drug-induced or radiation ILD/pneumonitis.
11. Immune-mediated rash from prior treatment that has not resolved prior to enrollment.
12. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 (with the exception of alopecia grade 2) at the time of starting study treatment.
13. Participant has concurrent or prior malignancy other than the disease under study. The following exceptions require consultation with the Medical Monitor:

    1. Non-muscle invasive bladder cancer (NMIBC) treated within the last 24 months that is considered completely cured. b. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured. c. Non-invasive cervical cancer treated within the last 24 months that is considered completely cured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion: an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Vailati Negrao, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org